CLINICAL TRIAL: NCT05243277
Title: Oculomotor Response While Using a Helmet Display Incorporating an Accommodation-vergence Stress Reduction Algorithm
Acronym: ALGO-HMD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PBMD04; 2021-A02286-35 (Other: IDRCB)
Record Dates: First submitted 2021-12-08; First posted 2022-02-17 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Visual Fatigue
Keywords: virtual reality
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Oculomotor tests — There will be four visits. Each visit is associated with a different exposure in terms of level of oculomotor conflict.
  At each visit, several oculomotor tests will be performed, followed by a comfort questionnaire. The oculomotor tests are subjective tests during which the participant will be asked to fix his/her eyes on one or more targets that can move in space and to indicate the way he/she perceives this/these target(s). Depending on the test, lenses may be inserted between the participant and the target to modify his/her perception.
  The comfort questionnaire consists to rate on a scale of 1 (not at all) to 5 (very much) the presence of visual symptoms, such as burning, watering or dryness.
  The participant will then have to perform four different perceptual tasks. His/her level of accommodation (i.e. focus) will be monitored throughout the tasks.
  Each exposure is followed again by eye tests and a comfort questionnaire.

SUMMARY:
Operational military personnel are increasingly using virtual or augmented reality headsets in the field or in training. However, these devices cause a conflict between accommodation (focus to see clearly) and vergence (alignment of both eyes on the object being viewed) that can be a source of visual fatigue and altered visual and perceptual abilities. Although techniques exist to limit this conflict for screen-based stimuli, the use of helmet visuals (or immersive headsets) adds technological complexity. Indeed, since accommodation on the screen of the helmet visual is impossible (i.e., distance too small) for the human visual system, lenses are used to virtually shift the image (referred to as a collimated image) so that accommodation can occur much further away. However, this material configuration also modifies the vergence, thus causing a conflict between accommodation and additional vergence that persists regardless of the attenuation technique used.

In this study, the investigator proposed to modify the image display to take into account the technical features of the helmet to correct this techno-dependent conflict. This study is aimed at determining whether the setting recommended by the algorithm developed by the investigator limits visual fatigue better than the conventional setting recommended by manufacturers or a subjective setting controlled by the user.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Non-presbyopic
* Stereoscopic acuity ≤ 60 min of arc

Exclusion Criteria:

* Accommodative insufficiency (APP ≤ 13-"age"/4, in diopters)
* Accommodative inertia (+ and - block in binocular)
* Compensation by orthokeratology
* Present or past binocular pathology: strabismus or amblyopia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is composed of healthy subjectfs with no history of visual disorders.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-12-16 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Evolution of oculomotor response to a stimulation generating jumps in vergence demand | Until the end of the study (20 months)
  Oculomotor response (accommodation and vergence) will be measured continuously via a single objective system (PowerRef 3) at each visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: Undecided